CLINICAL TRIAL: NCT02143505
Title: Calcium Plus Vitamin D Supplementation in Prevention of Colorectal Adenomas Recurrence:a Prospective, Randomized, Placebo-controlled, Multicenter Clinical Trial
Brief Title: Study of Calcium Plus Vitamin D Supplementation in Prevention of Colorectal Adenomas Recurrence
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Director of Department of Gastroenterology, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014BAI09B05
Record Dates: First submitted 2014-05-17; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Adenoma
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ca plus vit D (Experimental): elemental calcium 1200mg/d plus vitamin D3 250 IU/d daily supplements for 3 years
  Interventions: Drug: Ca plus vit D
- placebo (Placebo Comparator): identical-appearing placebo supplements for 3 years

INTERVENTIONS:
Drug: Ca plus vit D — elemental calcium 1200mg/d plus vitamin D3 250 IU/d daily supplements
  Other Names: Caltrate
  Arms: Ca plus vit D

SUMMARY:
Calcium plus vitamin D may be effective in the prevention of colorectal adenoma recurrence. The aim of this study is to investigate the effect of supplementation with calcium plus vitamin D on the recurrence of colorectal adenomas.

DETAILED DESCRIPTION:
Colorectal adenomas are well-known to be precancerous lesions that develop into colorectal cancers on the basis of the adenoma-carcinoma sequence. The effects of screening for colorectal adenomas and removing precancerous lesions on the prevention of colorectal cancer have been established. Because of the high recurrence rates of colorectal adenomas in patients who have undergone polypectomy, the potential chemopreventive agents that may reduce the risk of colorectal adenoma recurrence need to be investigated. Since laboratory and epidemiologic evidence suggests that calcium or vitamin D may help prevent colorectal adenomas, we conduct a randomized, placebo-controlled, prospective clinical trial to study the effect and safety of calcium plus vitamin D supplementation in prevention of colorectal adenomas recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65years
* Individuals who had at least one histologically confirmed colorectal adenoma removed within three months before recruitment
* Individuals without a history of familial polyposis
* Those who voluntarily sign the consent form after being fully informed and understanding the purpose and procedures of the study , characters of the disease, effect of medications, methods of related examinations, and potential risk/benefits of the study

Exclusion Criteria:

* Patients who are hypersensitive or intolerant to the drugs
* Patients who are intolerant to another colonoscopy examination
* Patients with hypercalcemia or urolithiasis
* Pregnant women, women during breast-feeding period, or women with expect pregnancy
* Patients with diabetes mellitus, severe heart or renal disease, or cancer history
* Patients with a history of subtotal gastrectomy or partial bowel resection
* Patients who are not able to cooperate
* Individual who are involved in designing, planning or performing this clinical trial
* Patients with medical conditions who are not appropriate to participate the study
* Patients who are taking aspirin, NSAIDs or COX2 inhibitors
* Patients who are taking folic acid or Butyrate.
* Patients with IBD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate recurrence rates of colorectal adenoma (CRA) after calcium plus vitamin D intervention. | 3 years

SECONDARY OUTCOMES:
The recurrence rates of advanced colorectal adenoma (A-CRA) after calcium plus vitamin D intervention. | 3 years

OTHER OUTCOMES:
changes in serum calcium | baseline and 3 years
changes in serum 25-(OH) Vit D level | baseline and 3 years
the incidence of colorectal cancer (CRC) after calcium plus vitamin D intervention | 3 years
changes in clinical symptoms scores (positive iFOBT, diarrhea, or constipation et al) | baseline and 3 years
differences in the number, location, size and histological subtype of CRA | baseline and 3 years
changes in routine blood count, urine and stool routine test, liver and kidney functions, etc | baseline and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yuan Fang, M.D., Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Institute of Digestive Disease, Shanghai, China